CLINICAL TRIAL: NCT05893641
Title: Investigate the Relationship Between Exercise Training and Recovery to Improve Physical Performance and Health Indices
Brief Title: Investigate the Relationship Between Exercise Training and Recovery Ratio to Improve Physical Performance and Health Status
Acronym: MOD_2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Gepner Yftach, Principal Investigator - Ph.D., Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0006524-1
Record Dates: First submitted 2023-05-09; First posted 2023-06-08 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Exercise; Recovery
Keywords: Recovery; Exercise training; Performance; Cardiometabolic health; Immune response
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A regular training volume (Active Comparator): They will maintain their training volume of 35 h/week
  Interventions: Behavioral: A regular training volume
- A lower exercise volume group (Active Comparator): They will conduct 85% of the control group weekly training volume (i.e., 30h/week)
  Interventions: Behavioral: A lower exercise volume group
- A longer rest group (Active Comparator): They will maintain the 35 h/week of exercise training, but with longer rest between exercise sessions
  Interventions: Behavioral: A longer rest group

INTERVENTIONS:
Behavioral: A regular training volume — Participate will maintain their training volume of 35 h/week
  Arms: A regular training volume
Behavioral: A lower exercise volume group — Participate will conduct 85% of the control group weekly training volume (i.e., 30h/week)
  Arms: A lower exercise volume group
Behavioral: A longer rest group — Participate will maintain the 35 h/week of exercise training
  Arms: A longer rest group

SUMMARY:
This study aims to investigate the effectiveness of various recovery strategies (such as longer recovery periods or reduced exercise intensity) in optimizing both physical performance and overall health status. Furthermore, the study will explore the potential of using changes in blood and urinary markers as indicators for assessing recovery status.

This study will assess whether extending recovery periods between exercise sessions and reducing the volume of exercise training can enhance the recovery process and enhance performance and health-related markers, relative to a control group.

One hundred-fifth young males will be recruited to participate in a single-center, parallel-group, randomized, well-controlled, superiority trial for 8 weeks of high-volume exercise training.

A single-center, parallel-group, randomized, well-controlled, superiority trial will be conducted among 150 physically active young males. Participants will undergo an 8-week high-volume exercise during base training program, which they will be randomly assigned to one of three groups: (1) a control group, which will follow the standard exercise regimen of 35 hours/week (n = 50); (2) a less exercise volume group, which will reduce exercise volume by 15% to 30 hours/week (n = 50); and (3) an extended recovery group, which will perform the same volume of exercise as the control group (35 hours/week), but with longer recovery intervals between exercises (n = 50). The intervention will take place at the Ministry of Defense training platform.

All study measurements will be taken at baseline and throughout the study. Body composition will be assessed using multichannel bioelectrical impedance (Seca). Continuously monitor (Garmin) will be used to evaluate heart rate and heart rate variability. Fasting blood samples will be used to examine inflammatory, lipid, glycemic, and endocrine markers. Physical performance will be assessed by several validated assessments, including handgrip, maximal voluntary contraction, Wingate test, Isometric Mid-Thigh Pull (IMTP), counter movement jump (CMJ) and maximal oxygen consumption (VO2max).

DETAILED DESCRIPTION:
The primary aim will be to determine the effect of different recovery strategies during 8 weeks of well-controlled, high-volume, large-scale, exercise training on the immune system (a), cardio-metabolic markers (b), and endocrine response (c).

Secondary aims will include: (1) To determine the effect of different recovery strategies during 8 weeks of well-controlled, high-volume, large-scale, exercise training on body strength (a), aerobic capacity (b), and body composition (c).

After baseline measurements, participants will be randomized 1:1:1 into one of three groups for 8 weeks: (1) a control group, which will follow the standard exercise regimen of 35 hours/week (n = 50); (2) a less exercise volume group, which will reduce exercise volume by 15% to 30 hours/week (n = 50); and (3) an extended recovery group, which will perform the same volume of exercise as the control group (35 hours/week), but with longer recovery intervals between exercises (n = 50).

Changes in health indices will be assessed by cardiometabolic, endocrine, and immune blood markers and body composition assessment at baseline (T0) after, 4 (T4), and 8 (T8) weeks of the intervention. Aerobic capacity, anaerobic threshold, and strength measurements will be used to determine changes in performance at T0, T4, and T8.

ELIGIBILITY:
Inclusion Criteria:

* Highly active participants
* Healthy
* Candidates for security course in the Ministry of Defense

Exclusion Criteria:

* Cardiopulmonary diseases (e.g., recent myocardial infarction or unstable angina)
* Musculoskeletal or neuromuscular impairments that preclude exercise training
* Cognitive impairments
* Use of drugs that affect bone or muscle metabolism (mainly steroids)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Changes in immune system | At baseline and at 8 weeks of intervention
  Tumor necrosis factor-a (pg/ml), Interleukin-6 (pg/ml)
Changes in immune system | At baseline and at 8 weeks of intervention
  C-Reactive protein (mg/dl)
Changes in cardiometabolic measurements | At baseline and at 8 weeks of intervention
  Glucose (mg/dl), lipid profile (total cholesterol in mg/dl, HDL in mg/dl, LDL in mg/dl)
Changes in endocrine measurements | At baseline and at 8 weeks of intervention
  Testosterone (ng/dL)
Changes in endocrine measurements | At baseline and at 8 weeks of intervention
  Growth hormone (ng/mL), Insulin-like growth factor 1 (ng/mL)

SECONDARY OUTCOMES:
Changes in aerobic capacity | At baseline and at 8 weeks of intervention
  Wingate test (watts)
Changes in aerobic capacity | At baseline and at 8 weeks of intervention
  Maximal O2 uptake (ml/kg/min)
Changes in body composition | At baseline and at 8 weeks of intervention
  BMI (kg/m^2)
Changes in body composition | At baseline and at 8 weeks of intervention
  waist circumference (cm)
Changes in body composition | At baseline and at 8 weeks of intervention
  Fat-free mass (kg)

OTHER OUTCOMES:
Changes in explosive power | At baseline and at 4 and 8 weeks of intervention
  Countermovement jump (in cm)
Strength assessment | At baseline and at 4 and 8 weeks of intervention
  Maximum voluntary contraction (in Newton)
Nutritional intake | At week 2 and week 6 of intervention
  protein intake (gr and in %of total kcal), carbohydrate intake (gr and in% of total kcal), fat intake (gr and in %of total kcal).
Nutritional intake | At week 2 and week 6 of intervention
  Will be assessed by validated questionnaires such as a food diary. Macronutrients composition will be measured from the self-reported nutritional intake: daily intake (kcal)

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Other, Israel

IPD SHARING:
Plan to Share IPD: No